CLINICAL TRIAL: NCT00034827
Title: A Multicenter Phase 2 Study of CI-1040 in Patients With Advanced Nonsmall-Cell Lung Cancer, Breast Cancer, Colon Cancer, or Pancreatic Cancer
Brief Title: A Multicenter Phase 2 Study of CI-1040 in Patients With Advanced Nonsmall-Cell Lung, Breast, Colon and Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1040-000-002
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2007-05-04 (Estimated); Status verified 2006-07

CONDITIONS: Colorectal Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms | interventions — 2-(2-chloro-4-iodophenylamino)-N-cyclopropylmethoxy-3,4-difluorobenzamide

INTERVENTIONS:
Drug: CI-1040

SUMMARY:
CI-1040 is an experimental drug that is being tested in patients who have advanced colorectal and lung cancer who failed no more than one prior chemotherapy regimen, breast cancer who have failed no more than 2 prior regimens and in patients with pancreatic cancer who have received no prior chemotherapy. CI-1040 is taken orally twice daily with meals. Patients are required to have blood tests periodically while receiving treatment and will be monitored closely throughout the trial for possible side effects and for response.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years or older who have pathological or hiostological confirmation of colorectal, nonsmall cell lung cancer, breast, or pancreas cancer.
* No more than 1 prior chemo for lung or colon cancer, no more than 2 for breast no prior chemotherapy for pancreas cancer.
* Original or recent tumor tissue must be available.
* Patients must have been off prior chemoptherapy for 4 weeks and radiation for 3 weeks.
* Patients must have adequate renal, liver, and bone marrow function, not have serious infection or life-threatening illness (unrelated to tumor).
* Must be able to swallow capsules and not have gastrointestinal disorders that may affect absorption of the drug.

Exclusion Criteria:

* Unstable medical condition
* prior chemotherapy within 4 week of screening
* series infection
* other tumor types
* ECOG performance status of 3 or 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172
Dates: Start 2002-01; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Overall objective response and clinical benefit response

SECONDARY OUTCOMES:
Time to objective response, duration of response, time to progression and survival

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (26):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Blendora, California
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Los Alamitos, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Mission Hills, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Oxnard, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Pomona, California
  - Pfizer Investigational Site, Rancho Cucamonga, California
  - Pfizer Investigational Site, Redondo Beach, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Ventura, California
  - Pfizer Investigational Site, West Covina, California
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, Cincinnait, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=1040-000-002&StudyName=A+Multicenter+Phase+2+Study+of+CI%2D1040+in+Patients+with+Advanced+Nonsmall%2DCell+Lung%2C+Breast%2C+Colon+and+Pancreatic+Cancer